CLINICAL TRIAL: NCT03458520
Title: Pediatric PET/MR Image Registry
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-44706; PEDSVAR0049 (Other: OnCore); 5U24CA264298-04 (NIH)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Soft Tissue; Lymphoma; Osteosarcoma
MeSH Terms: conditions — Lymphoma; Osteosarcoma | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Image Registry: patients with proven solid tumors or newly diagnosed mass strongly suspected to represent a solid tumor will receive MR imaging, PET/MR imaging (and if available, PET/CT imaging)
  Interventions: Diagnostic Test: PET/MR imaging; Diagnostic Test: MR imaging; Diagnostic Test: PET/CT imaging

INTERVENTIONS:
Diagnostic Test: PET/MR imaging — undergo PET/MR imaging
  Other Names: positron emission tomography
Diagnostic Test: MR imaging — Undergo MR imaging
  Other Names: magnetic resonance imaging
Diagnostic Test: PET/CT imaging — Undergo PET/CT imaging
  Other Names: computed tomography

SUMMARY:
The purpose of this study is to compare whole body magnetic resonance (MR) imaging, whole body positron emission tomography (PET)/MR imaging, and (if available) PET/Computed Tomography (CT) imaging for the diagnosis of tumors in children and young adults. Sensitivities, specificities and diagnostic accuracies of the different imaging modalities will be compared for significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients with proven solid tumors or newly diagnosed mass strongly suspected to represent a solid tumor.
* We might also include some patients with leukemia if there is concern for a focal lesion in any of their organs.
* Participant's parents (if participant is under 18) or the participant (if participant is 18 years or older) must willingly give written informed consent prior to any image transfer to the image registry.

Exclusion Criteria:

* Patient has contraindications for MRI or PET/MR. This includes patients with cardiac pacemakers or intracranial vascular clips as well as patients with a blood glucose level > 200 mg/dl.
* Lack of parental permission (if participant is younger than 18) or lack of informed consent (if participant is at least 18 years of age).
* Patient has a CNS primary tumor.
* Pregnant women and fetuses

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and young adult (<40 years) male or female subjects with proven solid tumors or newly diagnosed mass strongly suspected to represent a solid tumor
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of tumors | up to 12 months
  Number of tumors detected on whole body MRI, PET/MR and (if available) PET/CT scans.

SECONDARY OUTCOMES:
Metabolic activity of tumors | up to 12 months
  Metabolic activity of tumors determined by Standardized Uptake Values (SUV) on PET/MR and (if available) PET/CT scans.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Daldrup-Link, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States